CLINICAL TRIAL: NCT02807857
Title: A Prospective Evaluation of Natriuretic Peptide Based Referral of CHF Patients in Primary Care
Acronym: PREFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLCZ696B3402; 2016-000473-20 (EudraCT Number)
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Chronic Heart Failure (CHF)
Keywords: low-interventional observational study,; CHF,; heart failure,; primary care,; ESC guidelines,; Europe,; NT-proBNP,; reduced ventricular ejection fraction (EF),
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients' heart failure and non-heart failure (Other): No treatments are stipulated by this protocol - patients' HF and non-HF treatments will be observed throughout the study. The patients' treatment is entirely in the discretion of the primary care physicians
  Interventions: Procedure: Standard care

INTERVENTIONS:
Procedure: Standard care — Patients will receive the treatment that their primary care physician has decided to prescribe for their disease

SUMMARY:
This low interventional study, whose unique intervention was to measure the blood level of a biomarker called NT-proBNP in chronic heart failure patients daily followed-up by Primary Care Physicians (PCPs) in Europe, assessed if the cardiologist referral guided by NT-proBNP measurement in patients who were currently judged by PCPs as being stable, would lead to optimization of HF treatment, defined in adherence to treatment recommendations of the current European Society of Cardiology guidelines for the treatment of heart failure.

DETAILED DESCRIPTION:
In the majority of European countries, the primary management of chronic heart failure patients was performed by General Practitioners in collaboration with cardiologists (specialists). Previous studies had shown that many patients suffering from CHF do not receive optimal pharmacological and/or device treatment for their disease. An increase in natriuretic peptides (BNP, NT-proBNP) was associated with increased risk of cardiovascular events in heart failure patients. The purpose of the present study was to assess if a referral of clinical stable chronic heart failure patients with reduced ventricular ejection fraction (EF < or = 40%) and NT-proBNP level > or = 600 pg/mL to a specialist (cardiologist) led to treatment optimization, defined as adherence to the treatment recommendations according to the European Society of Cardiology (ESC) guidelines. In addition, data obtained in this study was used to describe demographic, clinical (including NT-proBNP levels) and treatment characteristics of CHF patients who were managed in the primary care setting across Europe..

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent and accept study procedures and time schedule.
* Age ≥ 18 years.
* Patients suffering from chronic heart failure (the heart failure diagnosis must have been made or confirmed by a cardiologist and/or hospital physician at any time in the patient's medical history).
* Patients with reduced ejection fraction (≤ 40%) as confirmed at any time point in the patient's medical history.

Exclusion Criteria:

* Use of investigational drugs either within 5 half-lives of enrollment, or within 30 days, or until the expected pharmacodynamic effect has returned to baseline, whichever is longer.
* Major surgery in the last 3 months prior to baseline or planned major surgery or cardiac intervention during the study.
* Cancer or other significant co-morbidities implying that the patient's condition is unstable.
* Comorbidities that can be associated with elevated natriuretic peptide (NP) levels: renal insufficiency, (eGFR < 25 ml/min/1.73 m² calculated according to MDRD formula), recent (less than 3 months) cerebral trauma or recent (less than 3 months) cerebrovascular incident, novel diagnosis or acute exacerbation of COPD within the last 3 months.
* Patients who are primarily managed and regularly followed-up by a cardiologist for their HF
* Highly frail patients whose estimated lifespan due to comorbidities by the judgement of the investigator is less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1415 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (167):
- Belgium (36):
  - Novartis Investigative Site, Kluisbergen, Belgium
  - Novartis Investigative Site, Binkom, BEL
  - Novartis Investigative Site, Gozée, BEL
  - Novartis Investigative Site, Linkebeek, BEL
  - Novartis Investigative Site, Oostham, BEL
  - Novartis Investigative Site, Zichem, BEL
  - Novartis Investigative Site, Aarschot
  - Novartis Investigative Site, Alveringem
  - Novartis Investigative Site, Boezinge
  - Novartis Investigative Site, Bruxe
  - Novartis Investigative Site, Buggenhout, Belgium
  - Novartis Investigative Site, Deinze
  - Novartis Investigative Site, Deurne
  - Novartis Investigative Site, Diksmuide
  - Novartis Investigative Site, Ezemaal-Neerwinden
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Hasselt, Belgium
  - Novartis Investigative Site, Herzele
  - Novartis Investigative Site, Landen
  - Novartis Investigative Site, Leefdaal
  - Novartis Investigative Site, Linkebeek
  - Novartis Investigative Site, Lommel
  - Novartis Investigative Site, Maasmechelen
  - Novartis Investigative Site, Mont-sur-Marchienne
  - Novartis Investigative Site, Nazareth
  - Novartis Investigative Site, Oosteeklo
  - Novartis Investigative Site, Ostend
  - Novartis Investigative Site, Oudenaarde
  - Novartis Investigative Site, Saint-Médard
  - Novartis Investigative Site, Stoumont
  - Novartis Investigative Site, Tessenderlo
  - Novartis Investigative Site, Thuilles
  - Novartis Investigative Site, Tielt-Winge
  - Novartis Investigative Site, Tremelo
  - Novartis Investigative Site, Vilvoorde
  - Novartis Investigative Site, Waregem
- Croatia (13):
  - Novartis Investigative Site, HRV, Croatia
  - Novartis Investigative Site, Rijeka, HRV
  - Novartis Investigative Site, Višnjevac, HRV
  - Novartis Investigative Site, Zagreb, HRV
  - Novartis Investigative Site, Bizovac
  - Novartis Investigative Site, HRV
  - Novartis Investigative Site, Krasica
  - Novartis Investigative Site, Osijek
  - Novartis Investigative Site, Rijeka
  - Novartis Investigative Site, Slavonski Brod
  - Novartis Investigative Site, Velika Kopanica
  - Novartis Investigative Site, Viškovo
  - Novartis Investigative Site, Zagreb
- Novartis Investigative Site, Nicosia, Cyprus
- Denmark (2):
  - Novartis Investigative Site, Præstø
  - Novartis Investigative Site, Skive
- Estonia (3):
  - Novartis Investigative Site, Sõmeru, EST
  - Novartis Investigative Site, Paide
  - Novartis Investigative Site, Tallinn
- France (19):
  - Novartis Investigative Site, Breteuil Sur Seine, France
  - Novartis Investigative Site, Arras
  - Novartis Investigative Site, Bersée
  - Novartis Investigative Site, Cannes
  - Novartis Investigative Site, Chantepie
  - Novartis Investigative Site, Colombiers
  - Novartis Investigative Site, Coursan
  - Novartis Investigative Site, Erquy
  - Novartis Investigative Site, La Seyne-sur-Mer
  - Novartis Investigative Site, Laval
  - Novartis Investigative Site, Les Pennes-Mirabeau
  - Novartis Investigative Site, Nègrepelisse
  - Novartis Investigative Site, Orthez
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rosiers d'Egleton
  - Novartis Investigative Site, Saint-Orens-de-Gameville
  - Novartis Investigative Site, Salles
  - Novartis Investigative Site, Six-Fours-les-Plages
  - Novartis Investigative Site, Strasbourg
- Hungary (15):
  - Novartis Investigative Site, Balatonkeresztúr
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Csongrád
  - Novartis Investigative Site, Érd
  - Novartis Investigative Site, Felsőrajk
  - Novartis Investigative Site, Hosszúhetény
  - Novartis Investigative Site, Kecskemét
  - Novartis Investigative Site, Korondi
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szabadsag
  - Novartis Investigative Site, Szeged-Szoreg
  - Novartis Investigative Site, Székesfehérvár
  - Novartis Investigative Site, Törökbálint
  - Novartis Investigative Site, Zákányszék
- Novartis Investigative Site, Beersheba, Israel
- Italy (2):
  - Novartis Investigative Site, Grumello del Monte, BG
  - Novartis Investigative Site, Gatteo, FC
- Latvia (3):
  - Novartis Investigative Site, Jelgava, LVA
  - Novartis Investigative Site, Riga, LVA
  - Novartis Investigative Site, Riga
- Lithuania (5):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Klaipėda, LTU
  - Novartis Investigative Site, Alytus
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Vilnius
- Malta (3):
  - Novartis Investigative Site, Xagħra, Gozo
  - Novartis Investigative Site, Xewkija, Gozo
  - Novartis Investigative Site, Rabat
- Norway (10):
  - Novartis Investigative Site, Ostereidet, Norway
  - Novartis Investigative Site, Flisa
  - Novartis Investigative Site, Hamar
  - Novartis Investigative Site, Hønefoss
  - Novartis Investigative Site, Kirkenær
  - Novartis Investigative Site, Lierskogen
  - Novartis Investigative Site, Lørenskog
  - Novartis Investigative Site, Løten
  - Novartis Investigative Site, Noetteroey
  - Novartis Investigative Site, Skien
- Poland (16):
  - Novartis Investigative Site, Chełm, POL
  - Novartis Investigative Site, Kartuzy, POL
  - Novartis Investigative Site, Warsaw, POL
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Bielawa
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Dzierżoniów
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Miasteczko Śląskie
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wieleń
  - Novartis Investigative Site, Wroclaw
  - Novartis Investigative Site, Zgierz
- Portugal (5):
  - Novartis Investigative Site, Seixal, Bairro Novo
  - Novartis Investigative Site, Cantanhede
  - Novartis Investigative Site, Leça da Palmeira
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Oeiras
- Russia (7):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Vladivostok
  - Novartis Investigative Site, Yaroslavl
- Slovenia (9):
  - Novartis Investigative Site, Ivančna Gorica
  - Novartis Investigative Site, Kranj
  - Novartis Investigative Site, Ljubljana
  - Novartis Investigative Site, Maribor
  - Novartis Investigative Site, Pesnica
  - Novartis Investigative Site, Slovenske Konjice
  - Novartis Investigative Site, Spodnji Duplek
  - Novartis Investigative Site, Vrhnika
  - Novartis Investigative Site, Žalec
- Spain (17):
  - Novartis Investigative Site, Cambre, A Coruna
  - Novartis Investigative Site, Porto do Son, A Coruña
  - Novartis Investigative Site, Petrel, Alicante
  - Novartis Investigative Site, El Parador de Las Hortichiuela, Almeria
  - Novartis Investigative Site, Alcúdia, Balearic Islands
  - Novartis Investigative Site, El Cañaveral, Caceres
  - Novartis Investigative Site, Puerto Real, Cadiz
  - Novartis Investigative Site, Burriana, Castellon
  - Novartis Investigative Site, Telde, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Parla, Madrid
  - Novartis Investigative Site, A Estrada, Pontevedra
  - Novartis Investigative Site, Monteporeiro, Pontevedra
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Panxón

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrolled set consisted of 1415 patients. 861 patients were referred to a cardiologist within this study and Based on findings from the interim-analysis, Novartis decided to terminate the study prematurely in March 2018.
Groups:
- Enrolled Patients: Adult male and female patients with chronic heart failure with reduced ejection fraction (LVEF ≤ 40%) who were managed in a primary care setting in sites across Europe. Patients who were considered clinically stable with NT-proBNP levels > 600 pg/ml were described and analyzed in the Follow-Up set.
Period: Enrolled Set
Arm/Group | Enrolled Patients
Started | 1415
Completed | 864
Not Completed | 551
Not completed — Patients not suitable for follow-up. | 551
Period: Follow-Up Set
Arm/Group | Enrolled Patients
Started | 864
Completed | 680
Not Completed | 184
Not completed — Study Terminated By Sponsor | 131
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 7
Not completed — Physician Decision | 6
Not completed — Adverse Event | 3
Not completed — Death | 27
Not completed — Relocation | 2

BASELINE CHARACTERISTICS:
Groups:
- Enrolled Patients: Adult male and female patients with chronic heart failure with reduced ejection fraction (LVEF ≤ 40%) who were managed in a primary care setting in sites across Europe. Patients who were considered clinically stable an with NT-proBNP levels > 600 pg/ml were referred to a cardiologist for evaluation and were in the follow-up set.
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 1415
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.8 (11.6)
Age, Customized [Number; unit: Participants] — Population: Enrolled Set
  Participants
    <65 years | 482
    ≥65 years to <75 years | 408
    ≥75 years to <85 years | 401
    ≥85 years | 124
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 436
  Male | 979
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1282
  More than one race | 0
  Unknown or Not Reported | 126

OUTCOME MEASURES:

1. Primary Outcome: Number of Clinically Stable Patients Whose Therapy Regimen Adheres to ESC Guideline Recommendations for Drug Types (Level 1) and Drug Type and Dose (Level 2) at Visit 1 (Before Referral to a Cardiologist)
Description: Assessment of treatment regimen with respect to ESC guideline adherence at Visit 1 before referral to cardiologist. ESC Criteria for adherence: Drug Types: Treatment with (1) ACEi or (1) ARB in combination with (1) beta-blocker and (1) MRA for patients w/an LVEF ≤ 35% at V1. Treatment w/(1) ACEi or (1) ARB, in combination with (1) beta-blocker+ without treatment with an MRA for patients with an LVEF > 35% at visit 1. Drug type & dose: Guideline adherent with respect to drug types and dosage of all respective guideline drugs ≥ 50% of the recommended target dose.
Time Frame: Baseline (Visit 1)
Population: Enrolled and Follow-up Set included. Due to missing left ventricular ejection fraction (LVEF) values, some patients could not be classified.
Measure: Number; unit: Participants
Groups:
- Enrolled Set: Adult male and female patients with chronic heart failure with reduced ejection fraction (LVEF ≤ 40%) who were managed in a primary care setting in sites across Europe.
- Follow-Up Set: Patients who were considered clinically stable and with NT-proBNP levels > 600 pg/ml who were referred to a cardiologist at Visit 1 for evaluation were in the follow-up set.
Arm/Group | Enrolled Set | Follow-Up Set
Number analyzed (Participants) | 1415 | 861
Participants
  Level 1: Drug Type : Adherent | 110 | 59
  Level 1: Drug type : Not Adherent | 802 | 523
  Patients missing LVEF values | 503 | 279

2. Primary Outcome: Adherence to ESC Guideline at Visit 2 (After Referral to a Cardiologist, Month 6), for Follow-up Set: Drug Type and Drug Type and Dose
Description: Assessment of patients' adherence at Visit 2, for patients who were already adherent at Visit 1, and those who were not adherent at Visit 1, for both drug type and drug type and dose. ESC Criteria for adherence: Drug Types: Treatment with (1) ACEi or (1) ARB in combination with (1) beta-blocker and (1) MRA for patients w/an LVEF ≤ 35% at V1. Treatment w/(1) ACEi or (1) ARB, in combination with (1) beta-blocker+ without treatment with an MRA for patients with an LVEF > 35% at visit 1. Drug type & dose: Guideline adherent with respect to drug types and dosage of all respective guideline drugs ≥ 50% of the recommended target dose.
Time Frame: Month 6
Population: Follow-Up set
Measure: Number; unit: Percentage of Patients
Arm/Group | Follow-Up Set
Number analyzed (Participants) | 861
Percentage of Patients
  Adherence at V2, not adherent at V1 for drug type | 3.3
  Adherence at V2, not adherent at V1:drug type/dose | 0.8
  Adherence at V2 and V1 for drug type | 79.2
  Adherence at Visit 1 for drug type & dose | 86.7

3. Secondary Outcome: Duration of Heart Failure
Description: The duration of Heart Failure was collected at Baseline (Visit 1).
Time Frame: Baseline (Visit 1)
Population: Enrolled Set and Follow-Up Set
Measure: Number; unit: Participants
Arm/Group | Enrolled Patients | Follow-Up Set
Number analyzed (Participants) | 1415 | 861
Participants
  >3 years | 896 | 549
  ≤3 years | 517 | 312

4. Secondary Outcome: Number of Patients With Current Use of Concomitant Compound
Description: Use of concomitant compounds were collected at baseline (Visit 1)
Time Frame: Baseline (Visit 1)
Population: Enrolled Set and Follow-Up Set
Measure: Number; unit: Participants
Arm/Group | Enrolled Set | Follow-Up Set
Number analyzed (Participants) | 1415 | 861
Participants
  Diuretics - without mineral corticoid antagonists | 934 | 625
  Beta blocking agents | 981 | 602
  Agents acting on the renin-angiotensin system | 834 | 491
  Diuretics - mineral corticoid antagonists | 664 | 416
  Antithrombotic agents | 401 | 256
  Cardiac therapy | 365 | 238
  Lipid modifying agents | 163 | 96
  Mineral supplements | 110 | 69
  Calcium channel blockers | 65 | 39

5. Secondary Outcome: Number of Follow-Up Patients With Current Use of Concomitant Compound at Visit 2
Description: Use of concomitant compounds were collected at 6 months (Visit 2)
Time Frame: 6 months (Visit 2)
Population: Follow-Up Set
Measure: Number; unit: Participants
Groups:
- Follow-Up Set Visit 2 (6 Months): Patients who were considered clinically stable and with NT-proBNP levels > 600 pg/ml were referred to a cardiologist after 6 months (V2) for evaluation and were in the follow-up set
Arm/Group | Follow-Up Set Visit 2 (6 Months)
Number analyzed (Participants) | 753
Participants
  Diuretics - without mineral corticoid antagonists | 581
  Beta blocking agents | 533
  Agents acting on the renin-angiotensin system | 476
  Diuretics - mineral corticoid antagonists | 423
  Antithrombotic agents | 221
  Cardiac therapy | 238
  Lipid modifying agents | 92
  Mineral supplements | 65
  Calcium channel blockers | 35

6. Secondary Outcome: Percentages of Clinically Stable Patients for Whom the Cardiologist and/or Primary Care Physician Optimizes Treatment Post Referral, Stratified According to Key Baseline Characteristics
Description: For patients who enter the prospective period of the study the post-referral treatment choice of cardiologists and/or primary care physicians was documented; for patients, for whom the cardiologist and/or primary care physician chose to prescribe a novel Heart Failure treatment, the treatment was assessed, if it fulfills the definition of adherence to European Society of Cardiology (ESC) guideline recommendation. The proportion of patients for whom an ESC guideline adherent treatment was de novo prescribed was assessed stratified according to different parameters.
Time Frame: 6 months
Population: Follow-Up Set
Measure: Number; unit: Percentage of Patients
Arm/Group | Follow-Up Set
Number analyzed (Participants) | 861
Percentage of Patients
  Cardiologist's advice-No change | 45.1
  Cardiologist's advice-Treatment intensification | 30.7
  Cardiologist's advice-Treatment reduction | 6.3
  Cardiologist's advice-Treatment adaption | 17.9

7. Secondary Outcome: Number of Patients With Different NT-proBNP Level Categories
Description: NT-proBNP levels (pg/ml) was measured at baseline in all consecutive patients who satisfy the inclusion and exclusion criteria. Measurements were performed on-site by means of a handheld device provided for the purposes of the study. NT-proBNP level categories could be 600 -799 pg/ml, 800 - 999 pg/ml, 1000 - 1200 pg/ml, > 1200 pg/ml).
Time Frame: One measurement in all consecutive patients at baseline (Visit 1)
Population: Enrolled Set and Follow-Up Set
Measure: Number; unit: Participants
Arm/Group | Enrolled Set | Follow-Up Set
Number analyzed (Participants) | 1415 | 861
Participants
  <600 pg/ml | 495 | 0
  ≥ 600 pg/ml to <800 pg/ml | 135 | 130
  ≥ 800 pg/ml to <1000 pg/ml | 97 | 93
  ≥ 1000 pg/ml to <1200 pg/ml | 80 | 75
  ≥ 1200 pg/ml to <1400 pg/ml | 48 | 46
  ≥ 1400 pg/ml to <1600 pg/ml | 32 | 24
  ≥ 1600 pg/ml to <1800 pg/ml | 33 | 33
  ≥ 1800 pg/ml to <2000 pg/ml | 30 | 29
  ≥ 2000 pg/ml | 465 | 431

8. Secondary Outcome: Percentages of Clinically Stable Patients
Description: Clinically stable patients in this study were defined as those patients for whom the primary care physician did not see a necessity (based on signs and symptoms of HF) to change the current pharmacological and/or device treatment of HF and who were on stable pharmacological and/or device treatment for HF for at least 3 months prior to inclusion.
Time Frame: Baseline (Visit 1)
Population: Enrolled Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Enrolled Set
Number analyzed (Participants) | 1415
Percentage of Participants
  Patients clinically stable | 96.9
  Patients not clinically stable | 3.1
  Patients suitable for prospective period of study | 63.2
  Patients not suitable for prospective period | 36.8

9. Secondary Outcome: Number of Patients by Cardiologist Prescription Practice Per Country/Region
Description: The cardiologists' suggestions for pharmacological and/or device therapy for the treatment of clinically stable CHF patients was documented and assessed by means of descriptive statistical measures stratified by country/region 6 months after baseline.
Time Frame: 6 months
Population: Follow-Up Set
Measure: Number; unit: Number of Participants
Arm/Group | Follow-Up Set
Number analyzed (Participants) | 861
Number of Participants
  Western EU | 198
  Eastern EU | 525

10. Secondary Outcome: Change of NT-proBNP Levels in Clinically Stable Chronic Heart Failure Patients With and Without Treatment Optimization 10 Months After Baseline
Description: At 10 months after baseline (end of study) NT-proBNP was assessed in clinically stable CHF patients with baseline NT-proBNP levels ≥ 600 pg/ml. Thus, for those patients two NT-proBNP measurements were available: at baseline and 10 months later. The individual change of NT-proBNP between both time points were assessed in accordance to the patients' treatment history during the study, i.e. baseline Heart Failure treatment and therapeutic decision taken 6 months after baseline.
Time Frame: 10 months
Population: Follow-Up Set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Follow-Up Set
Number analyzed (Participants) | 861
pg/mL
  NT-proBNP [pg/ml] at Visit 1 (Baseline) | 2753 (2530)
  NT-proBNP [pg/ml] at Visit 3 (10 months) | 2245 (2303)
  Absolute change in NT-proBNP (V3-V1) | -504 (2607)

11. Secondary Outcome: Change in EuroQol Five Dimensions Questionnaire (EQ-5D) Total and Individual Sub-scores at Visit 1 (Baseline), Visit 2 (6 Months) and Visit 3 (10 Months)
Description: Quality of life (QoL) was assessed by EQ-5D including the dimensions mobility, self-care, usual activity, pain/discomfort, anxiety/depression. A utility index based on UK value sets was built to summarize the information of these five dimensions into a single scale. The utility index can range between -0.281 and 1.0 where a higher number indicates a better health status. In addition, a visual analog scale (VAS) was applied with a possible range between 0 (=worst imaginable health state) and 100 (=best imaginable health state). Scores collected for all patients at baseline (Visit 1) and at Visit 2 and Visit 3 (only patients who entered the prospective period of the study, i.e. clinically stable patients with a NT-proBNP level ≥ 600 pg/ml) were asked to fill out the EuroQol 5D (EQ-5D) quality of life (QoL) questionnaire validated for heart failure (HF).
Time Frame: Baseline (Visit 1), 6 months (Visit 2), 10 months (Visit 3)
Population: Enrolled Set for Visit 1 (Baseline) and Follow-Up Set (Visit 2 and 3) for those clinically stable patients who entered the prospective period of the study
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Enrolled Set | Follow-Up Set
Number analyzed (Participants) | 1415 | 861
Scores on a scale
  EQ-5D Visual Analog Scale (VAS) - Visit 1: number analyzed (Participants) | 1411 | 860
  EQ-5D Visual Analog Scale (VAS) - Visit 1 | 60 [0 to 100] | 60 [0.0 to 100]
  EQ5D Utility index - Visit 1: number analyzed (Participants) | 1411 | 860
  EQ5D Utility index - Visit 1 | 0.81 [-0.17 to 1.00] | 0.79 [-0.17 to 1.00]
  EQ5D Utility index - Visit 2: number analyzed (Participants) | 0 | 747
  EQ5D Utility index - Visit 2 |  | 0.80 [-0.11 to 1.00]
  EQ5D Utility index absolute change (V2-V1): number analyzed (Participants) | 0 | 747
  EQ5D Utility index absolute change (V2-V1) |  | 0.00 [-0.47 to 0.83]
  EQ5D Utility index - Visit 3: number analyzed (Participants) | 0 | 569
  EQ5D Utility index - Visit 3 |  | 0.78 [0.28 to 1.00]
  EQ5D Utility index absolute change (V3-V1): number analyzed (Participants) | 0 | 567
  EQ5D Utility index absolute change (V3-V1) |  | 0.00 [-0.82 to 0.80]

12. Secondary Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Total and Individual Sub-scores at Visit 1 (Baseline), Visit 2 (6 Months) and Visit 3 (10 Months)
Description: The KCCQ is a self-administered questionnaire. It contains 23 items, covering physical function, clinical symptoms, social function, self-efficacy and knowledge, and quality of life, each with different Likert scale wording, including limitations, frequency, bother, change in condition, understanding, levels of enjoyment and satisfaction. Scores are transformed to a range of 0-100, in which higher scores reflect better health status. A positive change from baseline indicates improvement. Scores were collected for all patients at baseline and Visit 2 and Visit 3 (only patients who had entered the prospective period of the study (clinically stable patients with a NT-proBNP level ≥ 600 pg/ml) were asked to complete Kansas City Cardiomyopathy Questionnaire (KCCQ) validated for Heart Failure.
Time Frame: Baseline (Visit 1), 6 months (Visit 2), 10 months (Visit 3)
Population: as for outcome 11
Measure: Median (Full Range); unit: Utility Index Score
Arm/Group | Enrolled Set | Follow-Up Set
Number analyzed (Participants) | 1415 | 861
Utility Index Score
  KCCQ Total Symptom Score - Visit 1: number analyzed (Participants) | 1413 | 861
  KCCQ Total Symptom Score - Visit 1 | 77.1 [0 to 100] | 74.0 [0 to 100]
  KCCQ Clinical Summary Score - Visit 1: number analyzed (Participants) | 1413 | 861
  KCCQ Clinical Summary Score - Visit 1 | 72.1 [0 to 100] | 68.8 [0 to 100]
  KCCQ Overall Summary Score - Visit 1: number analyzed (Participants) | 1413 | 861
  KCCQ Overall Summary Score - Visit 1 | 70.1 [4.2 to 100] | 66.1 [4.2 to 100]
  KCCQ Overall Summary Score absolute change (V2-V1): number analyzed (Participants) | 0 | 747
  KCCQ Overall Summary Score absolute change (V2-V1) |  | 0.0 [-48.4 to 70.8]
  KCCQ Overall Summary Score - Visit 3: number analyzed (Participants) | 0 | 568
  KCCQ Overall Summary Score - Visit 3 |  | 66.7 [0.0 to 100]
  KCCQ Overall Summary Score absolute change (V3-V1): number analyzed (Participants) | 0 | 568
  KCCQ Overall Summary Score absolute change (V3-V1) |  | 0.5 [-66.1 to 66.8]
  KCCQ Clinical Summary Score - Visit 2: number analyzed (Participants) | 0 | 747
  KCCQ Clinical Summary Score - Visit 2 |  | 68.8 [1.0 to 100.0]
  KCCQ Clinical Summary Score abs. change (V2-V1): number analyzed (Participants) | 0 | 747
  KCCQ Clinical Summary Score abs. change (V2-V1) |  | 0.00 [-61.5 to 65.6]
  KCCQ Clinical Summary Score - Visit 3: number analyzed (Participants) | 0 | 568
  KCCQ Clinical Summary Score - Visit 3 |  | 68.8 [0.0 to 100.0]
  KCCQ Summary Score absolute change (V3-V1): number analyzed (Participants) | 0 | 568
  KCCQ Summary Score absolute change (V3-V1) |  | 0.0 [-53.1 to 69.0]

13. Secondary Outcome: Number of Patients in Different Living Conditions
Description: Living conditions were collected at Baseline (Visit 1).
Time Frame: Baseline (Visit 1)
Population: Enrolled Set and Follow-Up Set
Measure: Number; unit: Number of Participants
Arm/Group | Enrolled Set | Follow-Up Set
Number analyzed (Participants) | 1415 | 861
Number of Participants
  Living independently in household (alone) | 313 | 204
  Living with spouse or significant other | 817 | 481
  Living in residence with other family member | 264 | 159
  Living in a long term care facility | 20 | 16
  Transient housing | 1 | 1

14. Secondary Outcome: Number of Patients in Different Employment Status
Description: Employment status was collected at Baseline (Visit 1).
Time Frame: Baseline (Visit 1)
Population: Enrolled Set and Follow-Up Set
Measure: Number; unit: Number of Participants
Arm/Group | Enrolled Set | Follow-Up Set
Number analyzed (Participants) | 1415 | 861
Number of Participants
  Student | 0 | 0
  Employed (part-time) | 49 | 28
  Employed (full-time) | 144 | 51
  Homemaker | 26 | 15
  Retired | 1034 | 680
  Unemployed | 85 | 43
  Sustained Sick Leave | 73 | 40
  Missing | 4 | 4

15. Secondary Outcome: Number of Patients With Smoking Status
Description: Smoking status was collected at baseline (visit 1).
Time Frame: Baseline (Visit 1)
Population: Enrolled Set and Follow-Up Set
Measure: Number; unit: Number of Participants
Arm/Group | Enrolled Set | Follow-Up Set
Number analyzed (Participants) | 1415 | 861
Number of Participants
  Never | 779 | 500
  Current | 205 | 113
  Former | 427 | 246
  Missing | 4 | 2

16. Secondary Outcome: Number of Patients From Different Geographical Regions
Description: Geographic regions were collected at Baseline (Visit 1).
Time Frame: Baseline (visit 1)
Population: Enrolled Set
Measure: Number; unit: Number of Participants
Arm/Group | Enrolled Set | Follow-Up Set
Number analyzed (Participants) | 1415 | 861
Number of Participants
  RUS | 226 | 173
  BEL | 201 | 114
  HRV | 169 | 95
  SVN | 122 | 72
  POL | 120 | 74
  LTU | 103 | 65
  HUN | 94 | 58
  FRA | 89 | 54
  ESP | 76 | 30
  NOR | 58 | 33
  CYP | 36 | 20
  LVA | 34 | 22
  MLT | 26 | 17
  EST | 18 | 16
  DNK | 19 | 4
  PRT | 13 | 6

17. Secondary Outcome: Number of Patients With Health Insurance Status
Description: Health insurance status was collected at Baseline (Visit 1).
Time Frame: Baseline (Visit 1)
Population: Enrolled Set and Follow-Up Set
Measure: Number; unit: Number of Participants
Arm/Group | Enrolled Set | Follow-Up Set
Number analyzed (Participants) | 1415 | 861
Number of Participants
  Statutory Health Insurance | 1168 | 712
  Private Health Insurance | 29 | 22
  Combined statutory and private health insurance | 171 | 98
  None | 47 | 29

18. Secondary Outcome: Number of Patients at Different Educational Level
Description: Educational level was collected at Baseline (Visit 1).
Time Frame: Baseline (Visit 1)
Population: Enrolled Set and Follow-Up Set
Measure: Number; unit: Number of Participants
Arm/Group | Enrolled Set | Follow-Up Set
Number analyzed (Participants) | 1415 | 861
Number of Participants
  Primary Education | 396 | 248
  Secondary Education | 730 | 421
  University | 257 | 173
  None | 30 | 17
  Missing | 2 | 2

19. Secondary Outcome: Number of Patients Per Primary Etiology of Heart Failure
Description: The primary etiology of Heart Failure was collected at Baseline (Visit 1).
Time Frame: Baseline (Visit 1)
Population: Enrolled Set and Follow-Up Set
Measure: Number; unit: Number of Participants
Arm/Group | Enrolled Set | Follow-Up Set
Number analyzed (Participants) | 1415 | 861
Number of Participants
  Primary Etiology- Ischemic | 860 | 541
  Primary Etiology-Non-Ischemic | 553 | 320

20. Secondary Outcome: Number of Patients With Heart Failure (HF)-Related Hospitalizations in the Previous 12 Months Prior to Baseline, and During the Study
Description: HF-related hospitalizations was collected in the previous 12 months prior to baseline at baseline visit, at 6 and 10 months post-baseline.
Time Frame: Baseline (Visit 1), 6 months, 10 months
Population: Enrolled Set and Follow-Up Set
Measure: Number; unit: Number of Participants
Arm/Group | Enrolled Set | Follow-Up Set
Number analyzed (Participants) | 1415 | 861
Number of Participants
  Visit 1- Up to Baseline | 383 | 262
  Visit 2-6 months | 0 | 18
  Visit 3-10 months | 0 | 22
  Missing | 0 | 6

21. Secondary Outcome: Percentage of Patients With Cardiovascular and Non-cardiovascular Co-morbidities
Description: Cardiovascular and non-cardiovascular co-morbidities were collected at baseline (Visit 1)
Time Frame: Baseline (Visit 1)
Population: Enrolled Set and Follow-Up Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Enrolled Set | Follow-Up Set
Number analyzed (Participants) | 1415 | 861
Percentage of Participants
  Hypertension | 74.2 | 75.8
  Dyslipidemia | 61.6 | 58.8
  History of myocardial infarction | 43.9 | 44.4
  Atrial fibrillation | 40.8 | 52.3
  Obesity | 36.1 | 30.8
  Stable angina pectoris | 31.4 | 33.8
  Diabetes mellitus type 2 | 29.9 | 31.5
  Other Comorbidities | 13.0 | 14.0

22. Secondary Outcome: Mean Dose of Previously Taken and Current Use of Concomitant Medications
Description: Mean Dose of previously taken and current use of concomitant medications was to be collected at Visit 1, 6 months, 10 months post-baseline
Time Frame: Baseline (Visit 1), 6 months, 10 months
Population: Enrolled Set and Follow-Up Set (Mean dose of concomitant medications was not collected/provided and could not be alternately computed based upon the information listed).
Arm/Group | Enrolled Set | Follow-Up Set
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Number of Heart Failure (HF) Treatment Combinations
Description: The types and number of participants with HF treatment combinations were collected at Baseline (Visit 1).
Time Frame: Baseline (Visit 1)
Population: Follow-Up Set: Patients who were considered clinically stable and had NT-proBNP levels > 600 pg/ml who were referred to a cardiologist at Baseline (Visit 1) for evaluation.
Measure: Number; unit: Number of Participants
Arm/Group | Follow-Up Set
Number analyzed (Participants) | 861
Number of Participants
  One ACEi or one ARB and one beta-blocker(V1) | 178
  Exactly one beta-blocker and one MRA(V1) | 166
  Exactly one ACEi or one ARB and one MRA(V1) | 165
  One ACEi or (1)ARB & (1)MRA & (1)beta-blocker(V1) | 82
  Exactly one beta-blocker and ARNi(V1) | 13
  Exactly one MRA and ARNi(V1) | 20
  Exactly one MRA and one beta-blocker and ARNi(V1) | 9
  One ACEi or one ARB and one beta-blocker(V2) | 156
  Exactly one beta-blocker and one MRA(V2) | 160
  Exactly one ACEi or one ARB and one MRA(V2) | 177
  One ACEi or (1)ARB & (1)MRA & (1)beta-blocker(V2) | 91
  Exactly one beta-blocker and ARNi(V2) | 17
  Exactly one MRA and ARNi(V2) | 23
  Exactly one MRA and one beta-blocker and ARNi(V2) | 10
  One ACEi or one ARB and one beta-blocker(V3) | 120
  Exactly one beta-blocker and one MRA(V3) | 130
  Exactly one ACEi or one ARB and one MRA(V3) | 143
  One ACEi or (1)ARB & (1)MRA & (1)beta-blocker(V3) | 77
  Exactly one beta-blocker and ARNi(V3) | 11
  Exactly one MRA and ARNi(V3) | 17
  Exactly one MRA and one beta-blocker and ARNi(V3) | 6

24. Secondary Outcome: Duration of Treatment With Device Type
Description: The duration of treatment with device type was collected at baseline (Visit 1)
Time Frame: Baseline (Visit 1)
Population: Follow-Up Set (Data was not collected for this endpoint)
Arm/Group | Follow-Up Set
Number analyzed (Participants) | 0

25. Secondary Outcome: Duration of Previously Taken and Currently Use of Most Common Non-Heart Failure Concomitant Compounds
Description: Duration of most common previously taken and current use of most common Non-HF concomitant compounds were collected
Time Frame: Baseline (Visit 1)
Population: Follow-Up Set
Measure: Number; unit: Percentage of participants
Arm/Group | Follow-Up Set
Number analyzed (Participants) | 861
Percentage of participants
  Antithrombotic agents -≤1 and >3 years | 0.65
  Lipid modifying agents -≤1 and >3 years | 0.57
  Drugs for acid related disorders-≤1 and >3 years | 0.31

26. Secondary Outcome: Number of Patients by Primary Care Physicians' Prescription Practice Per Country/Region
Description: For clinically stable CHF patients, the primary care physicians' prescription of pharmacological and device treatment for HF was to be documented prior to baseline and post cardiologist-referral. At the post-referral visit the degree of implementation of cardiologist-recommendations and the medical decision making (e.g. reasons for non-implementation) were to be documented.
Time Frame: Baseline (Visit 1)
Population: Follow-Up Set (Data was not collected for this endpoint.)
Arm/Group | Follow-Up Set
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from FPFV to LPLV up to 2 years.
Arm/Group | Enrolled Set | Follow-Up Set
All-Cause Mortality (participants affected / at risk) | 32/1415 | 30/861
Serious Adverse Events (participants affected / at risk) | 117/1415 | 114/861
Other Adverse Events (participants affected / at risk) | 187/1415 | 181/861
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enrolled Set (N=1415) | Follow-Up Set (N=861)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Acute myocardial infarction (Cardiac disorders) | 3 | 3
Angina pectoris (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 9 | 9
Atrioventricular block (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 29 | 27
Cardiac failure acute (Cardiac disorders) | 2 | 2
Cardiac failure chronic (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 2
Myocardial infarction (Cardiac disorders) | 4 | 4
Palpitations (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 2 | 2
Melaena (Gastrointestinal disorders) | 1 | 1
Short-bowel syndrome (Gastrointestinal disorders) | 1 | 1
Chest discomfort (General disorders) | 1 | 1
Death (General disorders) | 3 | 2
Fatigue (General disorders) | 2 | 2
Oedema peripheral (General disorders) | 1 | 1
Soft tissue inflammation (General disorders) | 1 | 1
Sudden cardiac death (General disorders) | 1 | 1
Sudden death (General disorders) | 1 | 1
Ulcer haemorrhage (General disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Bacterial infection (Infections and infestations) | 1 | 1
Epididymitis (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Intestinal gangrene (Infections and infestations) | 1 | 1
Orchitis (Infections and infestations) | 1 | 1
Otitis externa (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 9 | 9
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 2
Electric shock (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 2 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1
International normalised ratio increased (Investigations) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 3
Fluid overload (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 4 | 4
Ischaemic stroke (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 5 | 5
Device malfunction (Product Issues) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 3
Renal failure (Renal and urinary disorders) | 1 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Homicide (Social circumstances) | 1 | 1
Aortic valve repair (Surgical and medical procedures) | 1 | 1
Cardiac ablation (Surgical and medical procedures) | 1 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 | 1
Cardiac resynchronisation therapy (Surgical and medical procedures) | 2 | 2
Cardioversion (Surgical and medical procedures) | 1 | 1
Circulatory collapse (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 1
Vasculitis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enrolled Set (N=1415) | Follow-Up Set (N=861)
Anaemia (Blood and lymphatic system disorders) | 6 | 6
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 5 | 5
Cardiac failure (Cardiac disorders) | 5 | 5
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Hypertensive cardiomyopathy (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 3 | 3
Tachyarrhythmia (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 6 | 6
Hypothyroidism (Endocrine disorders) | 1 | 1
Accommodation disorder (Eye disorders) | 1 | 1
Cataract (Eye disorders) | 4 | 4
Diplopia (Eye disorders) | 1 | 1
Sudden visual loss (Eye disorders) | 1 | 1
Visual acuity reduced (Eye disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 6
Dry mouth (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Enterocolitis (Gastrointestinal disorders) | 1 | 1
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 2 | 2
Gastroduodenitis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 2 | 2
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3
Adverse drug reaction (General disorders) | 1 | 1
Chest pain (General disorders) | 7 | 7
Fatigue (General disorders) | 9 | 9
Influenza like illness (General disorders) | 1 | 1
Localised oedema (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 8 | 8
Pyrexia (General disorders) | 1 | 1
Thirst (General disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 1
Bronchitis (Infections and infestations) | 10 | 10
Cellulitis (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Gingivitis (Infections and infestations) | 2 | 2
Influenza (Infections and infestations) | 2 | 2
Lower respiratory tract infection (Infections and infestations) | 2 | 2
Nasopharyngitis (Infections and infestations) | 4 | 4
Onychomycosis (Infections and infestations) | 1 | 1
Otitis media acute (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 2 | 2
Pulpitis dental (Infections and infestations) | 1 | 1
Pyuria (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 2 | 2
Skin infection (Infections and infestations) | 1 | 1
Tracheobronchitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 9 | 9
Viral infection (Infections and infestations) | 1 | 1
Viral sinusitis (Infections and infestations) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Blood creatinine abnormal (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 3 | 3
Blood iron decreased (Investigations) | 1 | 1
Blood pressure abnormal (Investigations) | 1 | 1
Blood pressure diastolic increased (Investigations) | 1 | 1
Haemoglobin increased (Investigations) | 1 | 1
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 1 | 1
Prostatic specific antigen increased (Investigations) | 1 | 1
Vitamin B12 decreased (Investigations) | 1 | 1
Weight decreased (Investigations) | 1 | 1
Weight increased (Investigations) | 2 | 2
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Obesity (Metabolism and nutrition disorders) | 3 | 3
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 8
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 3 | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 2
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 1
Cervical radiculopathy (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 5 | 5
Headache (Nervous system disorders) | 15 | 15
Hypoaesthesia (Nervous system disorders) | 1 | 1
Leukoencephalopathy (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 12 | 12
Anxiety disorder (Psychiatric disorders) | 2 | 2
Bipolar disorder (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 2 | 2
Hallucination, visual (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Nightmare (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 2 | 2
Nephropathy (Renal and urinary disorders) | 2 | 2
Nocturia (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 2
Renal colic (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 4 | 4
Urinary retention (Renal and urinary disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Blister (Skin and subcutaneous tissue disorders) | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Cataract operation (Surgical and medical procedures) | 2 | 2
Coronary angioplasty (Surgical and medical procedures) | 1 | 1
Dental operation (Surgical and medical procedures) | 1 | 1
Intraocular lens implant (Surgical and medical procedures) | 1 | 1
Aortic aneurysm (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 6 | 3
Hypotension (Vascular disorders) | 6 | 6
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 1 | 1
Varicose vein (Vascular disorders) | 1 | 1
Venous thrombosis (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
The recruitment was to be regarded as completed once approx. 2400 patients had entered the prospective period. However it was decided by Novartis to terminate the study prematurely, in March 2018.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-02-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT02807857/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT02807857/SAP_001.pdf